CLINICAL TRIAL: NCT06839495
Title: To Investigate the Relationship Between the Viscoelastic Properties of the Zona Pellucida of Human Oocyte and the Blastocyst Utilization Rate
Status: Recruiting | Type: Observational
Sponsor: Inti Labs (Industry)
Responsible Party: Sponsor
Other Study IDs: CS2-23192
Record Dates: First submitted 2025-02-13; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Oocyte; Zona Pellucida; Viscoelastic Property

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In in vitro fertilization (IVF) treatment, oocyte quality is one of the key factors influencing the success rate of fertilization. The zona pellucida (ZP) is a spherical structure that surrounds the human oocyte and, together with cumulus cells, forms the cumulus-oocyte complex (COC). These two components engage in bidirectional communication and metabolic regulation to support oocyte growth and maturation. Additionally, the physical rigidity of the zona pellucida plays an important role in the fertilization process.

OPAL X1 is a non-invasive and highly safe device specifically designed to measure the viscoelastic properties of the zona pellucida. This system consists of an ultra-precise pressure control mechanism and analytical software to assess oocyte quality before fertilization. OPAL X1 applies pressure through a micropipette while simultaneously recording the movement of the zona pellucida within the micropipette. An algorithm then analyzes the recorded motion images and classifies the oocytes into different quality grades (Grade A, B, C).

This study aims to investigate the correlation between oocyte classification results obtained from the OPAL X1 grading system and oocyte quality. By integrating spindle-view and time-lapse technology, the study seeks to identify the optimal parameters for oocyte quality assessment. Furthermore, these findings will be applied to predict the success rate of intracytoplasmic sperm injection (ICSI), the likelihood of blastocyst formation, and pregnancy outcomes after embryo transfer. Ultimately, this study aims to provide more efficient and timely embryo development information before IVF, assisting clinicians in formulating and optimizing IVF treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Women who have started the in vitro fertilization (IVF) treatment and related examinations.
2. Female participants aged ≤38 years with an anti-Müllerian hormone (AMH) concentration greater than 1.1 ng/mL and a collected oocyte count of more than 10.
3. Participants who consent to undergoing IVF with intracytoplasmic sperm injection (ICSI) and time-lapse embryo culture.

Exclusion Criteria:

1. Women diagnosed with untreated uterine abnormalities as assessed by a physician.
2. Participants with a body mass index (BMI) outside the range of 18.5-30 kg/m^2.
3. Patients undergoing IVF using sperm retrieved through surgical extraction.
4. Patients undergoing IVF using donated oocytes or donated sperm.

Max Age: 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women who have started the in vitro fertilization (IVF) treatment and related examinations.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Usable blastocyst rates | 4 weeks
  Usable blastocyst rates in each oocyte quality grading group.

SECONDARY OUTCOMES:
Pregnancy outcomes. | 12 months
  The correlation between oocyte quality grading groups and pregnancy outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Lee Women's Hospital, Taichung, Taiwan